CLINICAL TRIAL: NCT05323370
Title: Study of New Potential Biomarkers of Lymphangioleiomyomatosis: Determination of Cathepsin K, Cystatin C, Collagen Telopeptides and Chondroitin Sulfates
Brief Title: Lymphangioleiomyomatosis, a Study on Cathepsin K
Acronym: LAM-CAK
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR220020
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Lymphangioleiomyomatosis; Tuberous Sclerosis Complex
Keywords: urine
MeSH Terms: conditions — Lymphangioleiomyomatosis; Tuberous Sclerosis | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patientes with lymphangioleiomyomatosis: no intervention administered. Recruitment in pneumology department
  Interventions: Other: 24h urine; Other: urine sample
- Patientes with tuberous sclerosis complex without Lymphangioleiomyomatosis: no intervention administered. Recruitment in neurology department
  Interventions: Other: 24h urine; Other: urine sample
- Healthy women volunteers: no intervention administered. Recruitment in clinical investigation centre
  Interventions: Other: 24h urine; Other: urine sample

INTERVENTIONS:
Other: 24h urine — Urine samples will be collected at home over 24 hours
Other: urine sample — A urine sample of 20cc will be collected

SUMMARY:
This is a physiopathological case-control, non-interventional, monocentric study of adult patients with lymphangioleiomyomatosis. The controls are patients followed in neurology at the CHU of Tours for a tuberous sclerosis complex without lymphangioleiomyomatosis, the healthy volunteers are women with neither pulmonary nor renal pathology and recruited at the clinical investigation centre of the CHU of Tours.

ELIGIBILITY:
Inclusion criteria for patients with lymphangioleiomyomatosis

* Age ≥ 18 years
* Female carrier of lymphangioleiomyomatosis according to ERS criteria

Inclusion criteria for healthy female volunteers

* Age ≥ 18 years
* Women with no history of lymphangioleiomyomatosis, pulmonary, renal or osteoporotic disease

Inclusion criteria for tuberous sclerosis complex patients without lymphangioleiomyomatosis

* Age ≥ 18 years
* Woman followed for tuberous sclerosis complex for whom a chest CT scan less than 3 years old does not objectify a pulmonary cyst. (= without lymphangioleiomyomatosis)

Non-inclusion criteria

* Woman under judicial protection
* Woman with a urinary tract infection within 15 days
* Person who objected to the data processing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult female patients with lymphangioleiomyomatosis or with tuberous sclerosis complexwithout AML or healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
urine cathepsin K proteins levels | inclusion visit
  comparison of urine cathepsin K protein levels in the 3 groups
urine cathepsin K activity | inclusion visit
  comparison of urine cathepsin K activity in the 3 groups

SECONDARY OUTCOMES:
urinary quantity of cystatin C | inclusion visit
  comparison of urine cystacin C quantity in the 3 groups
urinary quantity C and N-telopeptides of type 1 collagen | inclusion visit
  comparison in the 3 groups
serum level of chondroitin sulphates | inclusion visit
  measurement in lymphangioleiomyomatosis patients
renal angiolipomas | inclusion visit
  measurement of the size of renal angiomyolipomas in lymphangioleiomyomatosis patients
FEV1 measurement | inclusion visit
  most recent FEV1 measurement as % of predicted value in lymphangioleiomyomatosis patients
VEGF-D measurement | inclusion visit
  most recent measurement of VEGF-D blood levels in lymphangioleiomyomatosis patients
T-score measurement | inclusion visit
  T-score measurement of the most recent bone densitometry in lymphangioleiomyomatosis patients

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain MARCHAND-ADAM, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided